CLINICAL TRIAL: NCT04550455
Title: A Prospective Biomarker Study in Active Secondary Progressive Multiple Sclerosis (SPMS)Subjects Treated With Cladribine Tablets
Brief Title: A Prospective Biomarker Study in Active SPMS Subjects Treated With Cladribine Tablets
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keith Edwards, M.D. (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor-Investigator, Keith Edwards, M.D., Director, Multiple Sclerosis Center of Northeastern New York
Organization: Multiple Sclerosis Center of Northeastern New York (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Cladribine-001
Record Dates: First submitted 2020-09-02; First posted 2020-09-16 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Intervention Model Description: Boxes for treatment cycles distributed will be based on weight
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cladribine Tablets (Experimental): All participants will receive cladribine tablets according to the current United States Federal Food and Drug Administration (FDA) package guidelines.
  Interventions: Drug: Cladribine Tablets

INTERVENTIONS:
Drug: Cladribine Tablets — Cladribine tablets will be administered according the current package insert guidelines
  Other Names: Mavenclad

SUMMARY:
The purpose of this study is to explore the concept that biomarker sensitivity will detect activity in Multiple Sclerosis (MS) subjects and allow appropriate change in treatment to prevent dysfunction.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a screening period. Maximum allowable time between first screening procedure and first administration of study treatment will be 42 days.

Subjects will have a 28 day run-in period consisting of 2 visits at week -4 and week -2.

Subjects will have a Baseline day 1 visit. Study medication will commerce on the day following this visit.

Additional visits will be at the following time points: week 4, week 8, week 12, week 16, week 24, week 36, week 48, week 52, week 56, week 60, week 72, week 84 and week 96.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 21 and 65 years old, inclusive.
2. Must be capable of understanding and providing written informed consent, including subject authorization under the health insurance portability and accountability act (HIPPA), prior to any study related procedures that are not part of routine medical care.
3. Has an EDSS score at the screening visit of 2.0 to 7.0 inclusive.
4. Have a diagnosis of clinically definite SPMS. (Lublin, 2014)
5. Are considered neurologically stable for > 30 days prior to both screening, baseline and week 48.
6. Must be otherwise healthy without confounding diseases.
7. Subject has decided to pursue cladribine tablets as their disease modifying therapy (DMT) of choice, and have signed a study specific informed consent form.
8. Must be willing and physically able to comply with all required protocol visits and complete all assessments.
9. Must be willing to complete 2 years of routine clinic follow-ups after study completion as per cladribine tablets FDA guidelines.
10. Must have read the FDA approved patient labeling (medication guide) and be counseled, risk of teratogenicity, lactation, lymphopenia and other hematologic toxicity, infections, liver injury, hypersensitivity, cardiac failure and treatment handling and administration.
11. If female: must have a negative serum pregnancy test at screen and week 48 and a negative urine pregnancy test at baseline. All females must agree to notify us immediately if they have concern of possible pregnancy.
12. If female: be neither pregnant or breastfeeding, nor attempting to conceive AND

    • Use a highly effective method of contraception throughout the entire duration of the study and for 6 months (5 menstrual cycles) following completion of the last dose of study medication. As it is currently unknown whether cladribine tablets may reduce the effectiveness of systemically acting hormonal contraceptives, a barrier method of contraception should be implemented for the duration of the study.
13. If Male: must be willing to use contraception to avoid contributing to pregnancies 6 months following the last dose of study medication.

Exclusion Criteria:

1. Subjects with a diagnosis of a sub-type of MS other than PMS active (clinically definite SPMS)
2. Have MRI findings other than MS that are considered significant per the P.I.
3. Have a clinical condition or medical history noted as a contraindication as per the FDA/US package insert guidelines.
4. Have a history of chronic disease(s) of the immune system, other than MS or a known immunodeficiency syndrome.
5. Have comorbid conditions that preclude participation, including any condition that might increase brain biomarkers such as traumatic brain injury (TBI), meningitis, stroke, or drug abuse in the last 12 months or any other medical condition deemed significant for increased biomarkers by the investigator.
6. Have an active/acute infection (bacterial, viral, fungal, etc.) at the time of screen AND/OR baseline or within 4 weeks prior to or at the start of course 2 year 2 that would interfere with the safety of the study.
7. Have a current or past significant history of poorly controlled diabetes mellitus, obesity (BMI over 35) or anorexia (BMI under 18), hypertension or hyperlipidemia as determined by the investigator.
8. Have a history or presence of malignancy other than basal cell epithelioma (BCE) or cervical cancer in-situ following a complete excision. Cancer that has been absent for more than 10 years and considered to be cured is allowed.

   a. All standard cancer screening guidelines should be followed for subjects that are treated with cladribine tablets during the course of the study.
9. Known liver conditions including the following:

   1. History or current hepatic impairment considered moderate or severe. Subjects with mild hepatic impairment can be considered at the investigator's discretion.
   2. Current or known history of alcohol abuse
   3. Chronic liver or biliary diseases
   4. Total or conjugated bilirubin greater than the upper limit of normal range
   5. Alkaline phosphatase (AP) greater than 1.5 times the upper limit of the normal range
   6. Aspartate transaminase (AST/ aka SGOT) and/or an alanine transaminase (ALT/aka SGPT) greater than 2 times the upper limit of normal range.
   7. Gamma-glutamyl-transferase (GGT) greater than 3 times the upper limit of normal.
10. History of or current renal Impairment that is considered moderate to severe. (creatinine clearance below 50 mL per minute)
11. Any other significant medical condition that in the opinion of the investigator that could potentially cause interference of complications of subject taking study Investigational Product (IP).
12. Have a contraindication to a lumbar puncture. (i.e. abnormal coagulation panel, skin infection at the location of Lumbar Puncture (LP), increased cranial pressure, etc.)
13. Any laboratory results at screen and/or prior to course 2 that are considered significant, such as but not limited to, abnormal lymphocyte count, positive hepatitis B and/or C screen, positive HIV test, etc. Any abnormal lab results must be approved by the investigator prior to initiating the first AND second course of IP therapy.
14. Have a lymphocyte count that is not at least 800 cells per microliter before initiating the second treatment course at week 48. If necessary, the second treatment course can be delayed as per FDA/US package insert guidelines.
15. Unable to undergo the required MRI scans for any reason, including claustrophobia and a history of hypersensitivity to Gd+.
16. Females who are pregnant, plan to become pregnant or who are breastfeeding during the study or plan on becoming pregnant or breastfeeding within 6 months of the last dose of cladribine tablets.
17. Males whose partner plans to become pregnant during the study or become pregnant within 6 months of the last dose of cladribine tablets.
18. Screening labs may be repeated in 2-6 weeks if an abnormality is felt to be due to a transient, reversible condition
19. Subjects that have previously been treated with cladribine in any dosing form (intravenous, subcutaneous, oral) are not allowed.
20. Subjects with a history of any of the following:

    1. Prior alemtuzumab treatment
    2. Prior or current investigational or non-FDA approved DMT or procedure
    3. Prior or current stem cell transplant for any reason
    4. Treatment with ocrelizumab or rituximab within 12 months of last dose to baseline
    5. Treatment with natalizumab within 1 year of screen. If subject has a prior history of treatment with natalizumab, the subject must also be JCV (John Cunningham virus) negative or have JCV index of 0.5 or lower. A past JCV index over 0.5 is exclusionary.
    6. Treatment with fingolimod, teriflunomide or dimethyl fumarate (DMF) within 4 weeks prior to baseline
    7. Treatment with interferon(IFN) or glatiramer acetate(GA) within 4 weeks of baseline
    8. Treatment with Intravenous immune globulin (IVIG) or plasmapheresis within 12 weeks prior to screening
    9. Treatment with an immunosuppressant such as cyclophosphamide, mitoxantrone, azathioprine, mycophenolate within 3 years prior to screening.
    10. Systemic corticosteroid within 2 weeks prior to screening. The screening period may be extended up to 4 weeks for patients who have used systemic corticosteroids but for a patient to be eligible for enrollment, no corticosteroids should be administered between screening and baseline
21. Treatment with concomitant drugs used for symptomatic treatment of spasticity or neuropathic pain, (i.e. baclofen, lorazepam, or gabapentin) as long as they have been stable dose for at least 30 days prior to screen. Medical Marijuana is allowed per investigator discretion and where allowed by state law. Medical Marijuana must not interfere with the subject's function.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to achieve no evidence of disease activity (NEDA) -4 compared to baseline | 96 weeks
  Currently accepted NEDA -3 criteria of 1) no clinical relapses 2) No new or newly enlarging MRI lesions 3) No progression of disability as measured by the expanded disability status scale (EDSS) with 4) the addition of no increase of serum and/or cerebrospinal fluid (CSF) and/or neurofilament light chain (NfL).
Decrease of serum/CSF NfL | 48 weeks
  Estimate of the change in serum/CSF NfL values from pre-treatment level to week 48

SECONDARY OUTCOMES:
Change in upper body function | 96 weeks
  Change in score, as recorded in seconds, measured by the 9- hole peg test. Lower Score is better
Change in Cognitive Function | 96 weeks
  Change in score as measured by the symbol digit modalities test (SDMT). Minimum Score =0 Maximum score =110. Higher Score is better

OTHER OUTCOMES:
CSF/serum glial fibrillary acidic protein (GFAP) | 96 weeks
  Values will be exploratory to determine if elevation of this value results in a meaningful change or stabilization over time
CSF/serum NfL antibody as markers for progressive multiple sclerosis (PMS) | 96 weeks
  Values will be exploratory to determine if elevation of this value results in a meaningful change or stabilization over time

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Edwards, M.D., Study Director — MS Center of Northeastern New York, P.C.
Locations (1):
- Multiple Sclerosis Center of Northeastern New York, P.C., Latham, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker D, Herrod SS, Alvarez-Gonzalez C, Zalewski L, Albor C, Schmierer K. Both cladribine and alemtuzumab may effect MS via B-cell depletion. Neurol Neuroimmunol Neuroinflamm. 2017 Jun 5;4(4):e360. doi: 10.1212/NXI.0000000000000360. eCollection 2017 Jul. PMID 28626781
- [Background] Bjornevik K, Munger KL, Cortese M, Barro C, Healy BC, Niebuhr DW, Scher AI, Kuhle J, Ascherio A. Serum Neurofilament Light Chain Levels in Patients With Presymptomatic Multiple Sclerosis. JAMA Neurol. 2020 Jan 1;77(1):58-64. doi: 10.1001/jamaneurol.2019.3238. PMID 31515562
- [Background] Brureau A, Blanchard-Bregeon V, Pech C, Hamon S, Chaillou P, Guillemot JC, Barneoud P, Bertrand P, Pradier L, Rooney T, Schussler N. NF-L in cerebrospinal fluid and serum is a biomarker of neuronal damage in an inducible mouse model of neurodegeneration. Neurobiol Dis. 2017 Aug;104:73-84. doi: 10.1016/j.nbd.2017.04.007. Epub 2017 Apr 6. PMID 28392472
- [Background] Comi G, Cook SD, Giovannoni G, Rammohan K, Rieckmann P, Sorensen PS, Vermersch P, Hamlett AC, Viglietta V, Greenberg SJ. MRI outcomes with cladribine tablets for multiple sclerosis in the CLARITY study. J Neurol. 2013 Apr;260(4):1136-46. doi: 10.1007/s00415-012-6775-0. Epub 2012 Dec 21. PMID 23263473
- [Background] Comi G, Cook S, Rammohan K, Soelberg Sorensen P, Vermersch P, Adeniji AK, Dangond F, Giovannoni G. Long-term effects of cladribine tablets on MRI activity outcomes in patients with relapsing-remitting multiple sclerosis: the CLARITY Extension study. Ther Adv Neurol Disord. 2018 Jan 23;11:1756285617753365. doi: 10.1177/1756285617753365. eCollection 2018. PMID 29399054
- [Background] Edwards KR, Garten L, Button J, O'Connor J, Kamath V, Frazier C. Neurofilament light chain as an indicator of exacerbation prior to clinical symptoms in multiple sclerosis. Mult Scler Relat Disord. 2019 Jun;31:59-61. doi: 10.1016/j.msard.2019.03.016. Epub 2019 Mar 23. PMID 30927733
- [Background] Freedman MS, Leist TP, Comi G, Cree BA, Coyle PK, Hartung HP, Vermersch P, Damian D, Dangond F. The efficacy of cladribine tablets in CIS patients retrospectively assigned the diagnosis of MS using modern criteria: Results from the ORACLE-MS study. Mult Scler J Exp Transl Clin. 2017 Oct 9;3(4):2055217317732802. doi: 10.1177/2055217317732802. eCollection 2017 Oct-Dec. PMID 29051829
- [Background] Feys P, Lamers I, Francis G, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. The Nine-Hole Peg Test as a manual dexterity performance measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):711-720. doi: 10.1177/1352458517690824. Epub 2017 Feb 16. PMID 28206826
- [Background] Gafson AR, Kim K, Cencioni MT, van Hecke W, Nicholas R, Baranzini SE, Matthews PM. Mononuclear cell transcriptome changes associated with dimethyl fumarate in MS. Neurol Neuroimmunol Neuroinflamm. 2018 Jun 12;5(4):e470. doi: 10.1212/NXI.0000000000000470. eCollection 2018 Jul. PMID 30283812
- [Background] Giovannoni G, Comi G, Cook S, Rammohan K, Rieckmann P, Soelberg Sorensen P, Vermersch P, Chang P, Hamlett A, Musch B, Greenberg SJ; CLARITY Study Group. A placebo-controlled trial of oral cladribine for relapsing multiple sclerosis. N Engl J Med. 2010 Feb 4;362(5):416-26. doi: 10.1056/NEJMoa0902533. Epub 2010 Jan 20. PMID 20089960
- [Background] Giovannoni G, Cook S, Rammohan K, Rieckmann P, Sorensen PS, Vermersch P, Hamlett A, Viglietta V, Greenberg S; CLARITY study group. Sustained disease-activity-free status in patients with relapsing-remitting multiple sclerosis treated with cladribine tablets in the CLARITY study: a post-hoc and subgroup analysis. Lancet Neurol. 2011 Apr;10(4):329-37. doi: 10.1016/S1474-4422(11)70023-0. PMID 21397565
- [Background] Giovannoni G, Cutter G, Sormani MP, Belachew S, Hyde R, Koendgen H, Knappertz V, Tomic D, Leppert D, Herndon R, Wheeler-Kingshott CAM, Ciccarelli O, Selwood D, di Cantogno EV, Ben-Amor AF, Matthews P, Carassiti D, Baker D, Schmierer K. Is multiple sclerosis a length-dependent central axonopathy? The case for therapeutic lag and the asynchronous progressive MS hypotheses. Mult Scler Relat Disord. 2017 Feb;12:70-78. doi: 10.1016/j.msard.2017.01.007. Epub 2017 Jan 17. PMID 28283111
- [Background] Giovannoni G, Soelberg Sorensen P, Cook S, Rammohan KW, Rieckmann P, Comi G, Dangond F, Hicking C, Vermersch P. Efficacy of Cladribine Tablets in high disease activity subgroups of patients with relapsing multiple sclerosis: A post hoc analysis of the CLARITY study. Mult Scler. 2019 May;25(6):819-827. doi: 10.1177/1352458518771875. Epub 2018 May 2. PMID 29716436
- [Background] Giovannoni G, Soelberg Sorensen P, Cook S, Rammohan K, Rieckmann P, Comi G, Dangond F, Adeniji AK, Vermersch P. Safety and efficacy of cladribine tablets in patients with relapsing-remitting multiple sclerosis: Results from the randomized extension trial of the CLARITY study. Mult Scler. 2018 Oct;24(12):1594-1604. doi: 10.1177/1352458517727603. Epub 2017 Sep 5. PMID 28870107
- [Background] Gold R, Giovannoni G, Selmaj K, Havrdova E, Montalban X, Radue EW, Stefoski D, Robinson R, Riester K, Rana J, Elkins J, O'Neill G; SELECT study investigators. Daclizumab high-yield process in relapsing-remitting multiple sclerosis (SELECT): a randomised, double-blind, placebo-controlled trial. Lancet. 2013 Jun 22;381(9884):2167-75. doi: 10.1016/S0140-6736(12)62190-4. Epub 2013 Apr 4. PMID 23562009
- [Background] Gregson A, Thompson K, Tsirka SE, Selwood DL. Emerging small-molecule treatments for multiple sclerosis: focus on B cells. F1000Res. 2019 Mar 1;8:F1000 Faculty Rev-245. doi: 10.12688/f1000research.16495.1. eCollection 2019. PMID 30863536
- [Background] Gunnarsson M, Malmestrom C, Axelsson M, Sundstrom P, Dahle C, Vrethem M, Olsson T, Piehl F, Norgren N, Rosengren L, Svenningsson A, Lycke J. Axonal damage in relapsing multiple sclerosis is markedly reduced by natalizumab. Ann Neurol. 2011 Jan;69(1):83-9. doi: 10.1002/ana.22247. Epub 2010 Dec 8. PMID 21280078
- [Background] Havrdova E, Galetta S, Hutchinson M, Stefoski D, Bates D, Polman CH, O'Connor PW, Giovannoni G, Phillips JT, Lublin FD, Pace A, Kim R, Hyde R. Effect of natalizumab on clinical and radiological disease activity in multiple sclerosis: a retrospective analysis of the Natalizumab Safety and Efficacy in Relapsing-Remitting Multiple Sclerosis (AFFIRM) study. Lancet Neurol. 2009 Mar;8(3):254-60. doi: 10.1016/S1474-4422(09)70021-3. Epub 2009 Feb 7. PMID 19201654
- [Background] Havrdova E, Arnold DL, Bar-Or A, Comi G, Hartung HP, Kappos L, Lublin F, Selmaj K, Traboulsee A, Belachew S, Bennett I, Buffels R, Garren H, Han J, Julian L, Napieralski J, Hauser SL, Giovannoni G. No evidence of disease activity (NEDA) analysis by epochs in patients with relapsing multiple sclerosis treated with ocrelizumab vs interferon beta-1a. Mult Scler J Exp Transl Clin. 2018 Mar 12;4(1):2055217318760642. doi: 10.1177/2055217318760642. eCollection 2018 Jan-Mar. PMID 29568544
- [Background] Hermann R, Karlsson MO, Novakovic AM, Terranova N, Fluck M, Munafo A. The Clinical Pharmacology of Cladribine Tablets for the Treatment of Relapsing Multiple Sclerosis. Clin Pharmacokinet. 2019 Mar;58(3):283-297. doi: 10.1007/s40262-018-0695-9. PMID 29987837
- [Background] Hogel H, Rissanen E, Barro C, Matilainen M, Nylund M, Kuhle J, Airas L. Serum glial fibrillary acidic protein correlates with multiple sclerosis disease severity. Mult Scler. 2020 Feb;26(2):210-219. doi: 10.1177/1352458518819380. Epub 2018 Dec 20. PMID 30570436
- [Background] Hutchinson M. The only certain measure of the effectiveness of multiple sclerosis therapy is cerebrospinal neurofilament level: Commentary. Mult Scler. 2015 Sep;21(10):1242-3. doi: 10.1177/1352458515599682. Epub 2015 Aug 4. No abstract available. PMID 26242693
- [Background] Kingwell E, Marriott JJ, Jette N, Pringsheim T, Makhani N, Morrow SA, Fisk JD, Evans C, Beland SG, Kulaga S, Dykeman J, Wolfson C, Koch MW, Marrie RA. Incidence and prevalence of multiple sclerosis in Europe: a systematic review. BMC Neurol. 2013 Sep 26;13:128. doi: 10.1186/1471-2377-13-128. PMID 24070256
- [Background] Kuhle J, Plavina T, Barro C, Disanto G, Sangurdekar D, Singh CM, de Moor C, Engle B, Kieseier BC, Fisher E, Kappos L, Rudick RA, Goyal J. Neurofilament light levels are associated with long-term outcomes in multiple sclerosis. Mult Scler. 2020 Nov;26(13):1691-1699. doi: 10.1177/1352458519885613. Epub 2019 Nov 4. PMID 31680621
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Leist TP, Comi G, Cree BA, Coyle PK, Freedman MS, Hartung HP, Vermersch P, Casset-Semanaz F, Scaramozza M; oral cladribine for early MS (ORACLE MS) Study Group. Effect of oral cladribine on time to conversion to clinically definite multiple sclerosis in patients with a first demyelinating event (ORACLE MS): a phase 3 randomised trial. Lancet Neurol. 2014 Mar;13(3):257-67. doi: 10.1016/S1474-4422(14)70005-5. Epub 2014 Feb 4. PMID 24502830
- [Background] Leppert D, Kuhle J. Serum NfL levels should be used to monitor multiple sclerosis evolution - Yes. Mult Scler. 2020 Jan;26(1):17-19. doi: 10.1177/1352458519872921. Epub 2019 Oct 18. No abstract available. PMID 31625807
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] Marrie RA, Goldman M. Validity of performance scales for disability assessment in multiple sclerosis. Mult Scler. 2007 Nov;13(9):1176-82. doi: 10.1177/1352458507078388. Epub 2007 Jul 10. PMID 17623733
- [Background] Noseworthy JH, Lucchinetti C, Rodriguez M, Weinshenker BG. Multiple sclerosis. N Engl J Med. 2000 Sep 28;343(13):938-52. doi: 10.1056/NEJM200009283431307. No abstract available. PMID 11006371
- [Background] Okai AF, Amezcua L, Berkovich RR, Chinea AR, Edwards KR, Steingo B, Walker A, Jacobs AK, Daizadeh N, Williams MJ; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ Investigators. Efficacy and Safety of Alemtuzumab in Patients of African Descent with Relapsing-Remitting Multiple Sclerosis: 8-Year Follow-up of CARE-MS I and II (TOPAZ Study). Neurol Ther. 2019 Dec;8(2):367-381. doi: 10.1007/s40120-019-00159-2. Epub 2019 Oct 25. PMID 31654272
- [Background] Pardo G, Jones DE. The sequence of disease-modifying therapies in relapsing multiple sclerosis: safety and immunologic considerations. J Neurol. 2017 Dec;264(12):2351-2374. doi: 10.1007/s00415-017-8594-9. Epub 2017 Sep 6. PMID 28879412
- [Background] Polman CH, O'Connor PW, Havrdova E, Hutchinson M, Kappos L, Miller DH, Phillips JT, Lublin FD, Giovannoni G, Wajgt A, Toal M, Lynn F, Panzara MA, Sandrock AW; AFFIRM Investigators. A randomized, placebo-controlled trial of natalizumab for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):899-910. doi: 10.1056/NEJMoa044397. PMID 16510744
- [Background] Przybek J, Gniatkowska I, Mirowska-Guzel D, Czlonkowska A. Evolution of diagnostic criteria for multiple sclerosis. Neurol Neurochir Pol. 2015;49(5):313-21. doi: 10.1016/j.pjnns.2015.07.006. Epub 2015 Aug 5. PMID 26377983
- [Background] Puentes F, van der Star BJ, Boomkamp SD, Kipp M, Boon L, Bosca I, Raffel J, Gnanapavan S, van der Valk P, Stephenson J, Barnett SC, Baker D, Amor S. Neurofilament light as an immune target for pathogenic antibodies. Immunology. 2017 Dec;152(4):580-588. doi: 10.1111/imm.12797. Epub 2017 Aug 11. PMID 28718500
- [Background] Rochwerg B, Almenawer SA, Siemieniuk RAC, Vandvik PO, Agoritsas T, Lytvyn L, Alhazzani W, Archambault P, D'Aragon F, Farhoumand PD, Guyatt G, Laake JH, Beltran-Arroyave C, McCredie V, Price A, Chabot C, Zervakis T, Badhiwala J, St-Onge M, Szczeklik W, Moller MH, Lamontagne F. Atraumatic (pencil-point) versus conventional needles for lumbar puncture: a clinical practice guideline. BMJ. 2018 May 22;361:k1920. doi: 10.1136/bmj.k1920. No abstract available. PMID 29789372
- [Background] Rudick RA, Stuart WH, Calabresi PA, Confavreux C, Galetta SL, Radue EW, Lublin FD, Weinstock-Guttman B, Wynn DR, Lynn F, Panzara MA, Sandrock AW; SENTINEL Investigators. Natalizumab plus interferon beta-1a for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):911-23. doi: 10.1056/NEJMoa044396. PMID 16510745
- [Background] SCHUMACHER GA, BEEBE G, KIBLER RF, KURLAND LT, KURTZKE JF, MCDOWELL F, NAGLER B, SIBLEY WA, TOURTELLOTTE WW, WILLMON TL. PROBLEMS OF EXPERIMENTAL TRIALS OF THERAPY IN MULTIPLE SCLEROSIS: REPORT BY THE PANEL ON THE EVALUATION OF EXPERIMENTAL TRIALS OF THERAPY IN MULTIPLE SCLEROSIS. Ann N Y Acad Sci. 1965 Mar 31;122:552-68. doi: 10.1111/j.1749-6632.1965.tb20235.x. No abstract available. PMID 14313512
- [Background] Schwartz CE, Powell VE. The Performance Scales disability measure for multiple sclerosis: use and sensitivity to clinically important differences. Health Qual Life Outcomes. 2017 Mar 9;15(1):47. doi: 10.1186/s12955-017-0614-z. PMID 28274258
- [Background] Stankiewicz JM, Weiner HL. An argument for broad use of high efficacy treatments in early multiple sclerosis. Neurol Neuroimmunol Neuroinflamm. 2019 Nov 22;7(1):e636. doi: 10.1212/NXI.0000000000000636. Print 2020 Jan. PMID 31757815
- [Background] Strober L, DeLuca J, Benedict RH, Jacobs A, Cohen JA, Chiaravalloti N, Hudson LD, Rudick RA, LaRocca NG; Multiple Sclerosis Outcome Assessments Consortium (MSOAC). Symbol Digit Modalities Test: A valid clinical trial endpoint for measuring cognition in multiple sclerosis. Mult Scler. 2019 Nov;25(13):1781-1790. doi: 10.1177/1352458518808204. Epub 2018 Oct 18. PMID 30334474
- [Background] Scalfari A, Knappertz V, Cutter G, Goodin DS, Ashton R, Ebers GC. Mortality in patients with multiple sclerosis. Neurology. 2013 Jul 9;81(2):184-92. doi: 10.1212/WNL.0b013e31829a3388. PMID 23836941
- [Background] Trapp BD, Peterson J, Ransohoff RM, Rudick R, Mork S, Bo L. Axonal transection in the lesions of multiple sclerosis. N Engl J Med. 1998 Jan 29;338(5):278-85. doi: 10.1056/NEJM199801293380502. PMID 9445407
- [Background] Montalban X, Gold R, Thompson AJ, Otero-Romero S, Amato MP, Chandraratna D, Clanet M, Comi G, Derfuss T, Fazekas F, Hartung HP, Havrdova E, Hemmer B, Kappos L, Liblau R, Lubetzki C, Marcus E, Miller DH, Olsson T, Pilling S, Selmaj K, Siva A, Sorensen PS, Sormani MP, Thalheim C, Wiendl H, Zipp F. ECTRIMS/EAN Guideline on the pharmacological treatment of people with multiple sclerosis. Mult Scler. 2018 Feb;24(2):96-120. doi: 10.1177/1352458517751049. Epub 2018 Jan 20. PMID 29353550
- [Background] Nielsen AS, Kinkel RP, Madigan N, Tinelli E, Benner T, Mainero C. Contribution of cortical lesion subtypes at 7T MRI to physical and cognitive performance in MS. Neurology. 2013 Aug 13;81(7):641-9. doi: 10.1212/WNL.0b013e3182a08ce8. Epub 2013 Jul 17. PMID 23864311
- [Background] Kollia K, Maderwald S, Putzki N, Schlamann M, Theysohn JM, Kraff O, Ladd ME, Forsting M, Wanke I. First clinical study on ultra-high-field MR imaging in patients with multiple sclerosis: comparison of 1.5T and 7T. AJNR Am J Neuroradiol. 2009 Apr;30(4):699-702. doi: 10.3174/ajnr.A1434. Epub 2009 Jan 15. PMID 19147714
- [Background] Pitt D, Boster A, Pei W, Wohleb E, Jasne A, Zachariah CR, Rammohan K, Knopp MV, Schmalbrock P. Imaging cortical lesions in multiple sclerosis with ultra-high-field magnetic resonance imaging. Arch Neurol. 2010 Jul;67(7):812-8. doi: 10.1001/archneurol.2010.148. PMID 20625086
- [Background] Kister I, Bacon TE, Chamot E, Salter AR, Cutter GR, Kalina JT, Herbert J. Natural history of multiple sclerosis symptoms. Int J MS Care. 2013 Fall;15(3):146-58. doi: 10.7224/1537-2073.2012-053. PMID 24453777
- [Background] Salter A, Thomas N, Tyry T, Cutter G, Marrie RA. Employment and absenteeism in working-age persons with multiple sclerosis. J Med Econ. 2017 May;20(5):493-502. doi: 10.1080/13696998.2016.1277229. Epub 2017 Jan 25. PMID 28035846
- [Background] Correale J, Gaitan MI, Ysrraelit MC, Fiol MP. Progressive multiple sclerosis: from pathogenic mechanisms to treatment. Brain. 2017 Mar 1;140(3):527-546. doi: 10.1093/brain/aww258. PMID 27794524
- [Background] Confavreux C, Vukusic S, Moreau T, Adeleine P. Relapses and progression of disability in multiple sclerosis. N Engl J Med. 2000 Nov 16;343(20):1430-8. doi: 10.1056/NEJM200011163432001. PMID 11078767
- [Background] Jack D, Nolting A, Galazka A. Favorable outcomes after COVID-19 infection in multiple sclerosis patients treated with cladribine tablets. Mult Scler Relat Disord. 2020 Nov;46:102469. doi: 10.1016/j.msard.2020.102469. Epub 2020 Aug 27. No abstract available. PMID 32919180
- See also: Protocol Reference # 7 — https://onlinelibrary.ectrims-congress.eu/ectrims/2016/32nd/146475/s.cook.cladribine.tablets.in.the.treatment.of.patients.with.multiple.sclerosis.html?f=listing%3D0%2Abrowseby%3D8%2Asortby%3D1%2Asearch%3Dcladribine+tablets%2Btreatment%2Bpatients%2Bmultiple+sclerosis%3A%2Bintegrated+analysis
- See also: Protocol Reference # 9 — https://apps.who.int/iris/handle/10665/43968
- See also: Protocol Reference #12 — https://www.emdserono.com/us-en/pi/mavenclad-mg.pdf
- See also: Protocol Reference # 14 — https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/022561s000lbl.pdf
- See also: Protocol Reference # 22 — https://onlinelibrary.ectrims-congress.eu/ectrims/2016/32nd/146476/gavin.giovannoni.benefits.of.cladribine.tablets.on.the.proportion.of.patients.html?f=listing%3D0%2Abrowseby%3D8%2Asortby%3D1%2Asearch%3Dbenefits%2Bcladribine+tablets%2Bproportion%2Bpatients%2Bmultiple+sclerosis+free%2Bclinical%2Bradiological
- See also: Protocol Reference #55 — https://onlinelibrary.ectrims-congress.eu/ectrims/2017/ACTRIMS-ECTRIMS2017/199999/mitchell.t.wallin.the.prevalence.of.multiple.sclerosis.in.the.united.states.a.html
- See also: Protocol Reference # 61 — https://files.eric.ed.gov/fulltext/ED444296.pdf